CLINICAL TRIAL: NCT07124481
Title: Early Mindfulness Based Cognitive Therapy for Prevention of Psychological Distress in Cancer Patients
Acronym: EarlyMind
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Collaborators: Helen Dowling Institute (Unknown)
Responsible Party: Principal Investigator, Marit Mentink, PhD, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2306
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Mindfulness Based Cognitive Therapy
MeSH Terms: conditions — Neoplasms | interventions — Mindfulness-Based Stress Reduction; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): mindfulness based stress reduction
  Interventions: Behavioral: Mindfulness based stress reduction
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — 8 weekly sessions of 2.5 hour per session, face-to-face in a group consisting of maximum 15 participants, supervised by a certified mindfulness trainer
  Other Names: mindfulness; mindfulness therapy; MBCT
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if early provision of mindfulness based cognitive therapy can prevent psychological distress in adult patients with cancer one year after diagnosis.

Researchers will compare mindfulness based cognitive therapy to usual care to see if psychological distress is lower in patients that followed mindfulness.

Participants will follow 8 weekly sessions of mindfulness and fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with urological cancer or breast cancer
* <6 weeks since cancer diagnosis
* Planned curative treatment or palliative treatment with life expectation >1 year
* Good proficiency in Dutch language

Exclusion Criteria:

* Serious psychiatric history or current psychiatric treatment (interfering with study participation): 1) current suicidal ideation, 2) current psychosis or bipolar disorder, 3) psychosis or bipolar disorder in history
* Unable to understand study procedure
* A priori unable to be available for 8 week MBCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Psychological distress | From enrollment to 2 years after diagnosis
  Anxiety and depression as measured with the Hospital Anxiety and Depression Scale

IPD SHARING:
Plan to Share IPD: Undecided